CLINICAL TRIAL: NCT07234838
Title: Influence of Anti-Psoriatic Biologic Therapies Targeting TNF-α and Interleukins 17 and 23 on the Risk of Development and Recurrence of Anogenital Warts: A Retrospective and Prospective Study With an Exploratory Component on HPV Vaccination Acceptability (CONDYPSO)
Brief Title: Effect of Anti-Psoriatic Biologics on Risk of Anogenital Warts (CONDYPSO)
Acronym: CONDYPSO
Status: Not yet recruiting | Type: Observational
Sponsor: Jonathan Krygier (Other)
Responsible Party: Sponsor-Investigator, Jonathan Krygier, Dr, Centre Hospitalier Universitaire Saint Pierre
Organization: Centre Hospitalier Universitaire Saint Pierre (Other)
Other Study IDs: HUB2025494; 1st Medical Council Grant (Other Grant/Funding Number: Association for Medical Research Support André Vésale (non-profit association))
Record Dates: First submitted 2025-10-02; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis; Condyloma Acuminata; Biotherapies
Keywords: psoriasis; Influence of Anti-Psoriatic Biologic Therapies; Risk of Development and Recurrence of Anogenital Warts
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — curettage specimen of anogenital warts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Biologic therapies (Anti-TNF, Anti-IL-17, Anti-IL-23, including ustekinumab): Psoriasis patients receiving biologic therapies. Observational follow-up of anogenital HPV-related outcomes (warts, recurrences, cytology, vaccination acceptability).
- Other immunomodulators (methotrexate, cyclosporine, deucravacitinib, dimethyl fumarate): Psoriasis patients receiving systemic immunomodulators other than biologics. Observational follow-up of anogenital HPV-related outcomes.
- Other systemic non-immunomodulators (apremilast, acitretin): Psoriasis patients receiving systemic therapies not primarily immunomodulatory. Observational follow-up of anogenital HPV-related outcomes.
- Topical therapy only (topical corticosteroids, calcineurin inhibitors, phototherapy): Psoriasis patients managed with topical therapy and/or phototherapy only. Observational follow-up of anogenital HPV-related outcomes.
- Untreated psoriasis patients: Psoriasis patients currently not receiving any systemic or topical therapy. Observational follow-up of anogenital HPV-related outcomes.

SUMMARY:
This study aims to assess the impact of anti-TNF-α, anti-IL-17, and anti-IL-23 biologic therapies on the risk of development or recurrence of anogenital warts (AGW) in patients with moderate to severe psoriasis. By modulating systemic and mucosal immunity, these treatments may alter host defenses against human papillomavirus (HPV) infections, which are responsible for AGW. In particular, inhibition of Th1 pathways (by anti-TNF-α) and Th17 pathways (by anti-IL-17 and anti-IL-23), both central to the antiviral response, may reduce local production of pro-inflammatory cytokines (such as IFN-γ, IL-17, and IL-22), decrease the activity of CD8+ cytotoxic T lymphocytes, and impair dendritic cell function, thereby compromising viral clearance at the genital mucosa.

AGW are a frequent and recurrent manifestation of HPV infection, and their incidence may be influenced by these immunomodulatory treatments.

The retrospective component will review cases already documented in medical records and analyze, to the extent permitted by available data, the same risk factors as in the prospective component, including history of sexually transmitted infections (STIs), risk behaviors, treatments used (systemic or topical), and time to onset or recurrence of AGW. This analysis will be conducted as a retrospective case-control study, matching each patient who developed AGW with one or more controls receiving biologics who did not develop AGW, in order to identify factors associated with their occurrence.

The prospective follow-up will assess, over 24 months, risk factors for occurrence or recurrence of AGW in patients with moderate to severe psoriasis, according to the treatment received: no treatment, topical treatment, systemic non-immunomodulatory treatment, or immunomodulatory treatment, including biologics. Acceptability of HPV vaccination will also be evaluated in this adult population treated with immunomodulators, which remains insufficiently targeted by current vaccination recommendations.

DETAILED DESCRIPTION:
Scientific Rationale

Anogenital warts (AGW) are a frequent manifestation of human papillomavirus (HPV) infection. Their course is generally benign, but they may cause significant discomfort and carry a high risk of recurrence, particularly in the context of immunomodulation.

Psoriasis is a chronic inflammatory skin disease affecting approximately 2-3% of the global population. Biologic therapies targeting IL-17 and IL-23, now widely used, profoundly modulate mucosal immunity by acting on the Th17 axis. This pathway plays a central role in defense against viral and fungal pathogens on mucosal surfaces, notably through the production of IL-17 and IL-22. Their inhibition leads to a decrease in these cytokines, which could theoretically impair local viral clearance, particularly with respect to HPV, thereby promoting persistence or recurrence of AGW.

Anti-TNF-α agents, long used in dermatology, also influence antiviral immunity by reducing the activity of cytotoxic CD8+ T lymphocytes and the production of IFN-γ, a key Th1 cytokine.

This rationale is supported by experimental data showing the essential role of Th1 and Th17 pathways, CD8+ lymphocytes, dendritic cells, and IFN-γ in the control of HPV infections.

A cross-sectional study in 222 patients with psoriasis or inflammatory bowel disease, including 104 treated with anti-TNF-α, did not demonstrate a significant increase in the prevalence of anogenital HPV infections compared with patients receiving alternative therapies or no treatment. At baseline, the analysis combined grouped anogenital swabs (penis or vulva, perianal area, and cervix in women) with broad-spectrum HPV PCR, together with serology for neutralizing antibodies against genotypes 6, 16, and 18. However, this study does not allow conclusions on the long-term safety of these treatments, nor on the risk associated with individual molecules, due to sample size and the cross-sectional design.

Another, more recent cross-sectional study suggested an increased prevalence of oral HPV infections in psoriatic patients treated for at least 6 months with anti-IL-17, particularly after prolonged exposure (>8 years), compared with patients receiving topical treatments or other biologics (anti-TNF-α or ustekinumab). HPV PCR on oral rinse was performed at a single time point at inclusion. Genital infections were also investigated using perineal swabs with PCR analysis, but results were less conclusive, with no statistically significant differences between groups.

Several case reports have described the occurrence or worsening of AGW in patients receiving anti-IL-17 or anti-TNF-α, suggesting a possible negative impact on viral clearance. These remain isolated observations and do not establish causality.

Conversely, elevated levels of interleukins 17 and 23 have been detected in HPV-induced lesions, particularly in the cervix and anal canal. Their inhibition might therefore exert a protective effect against the progression of HPV-induced lesions.

Cases of regression of warts, including AGW and cutaneous warts, have indeed been reported under anti-IL-17, as well as a case of regression of high-grade HPV-associated dysplasia after switching from an anti-IL-12/23 (ustekinumab) to a selective anti-IL-23 (risankizumab). To date, no cases of AGW have been reported with the newer anti-IL-23 agents such as guselkumab, risankizumab, or tildrakizumab, while a single isolated case under ustekinumab was published in 2021.

A review of the literature confirms the lack of robust quantitative data in patients treated with IL-17 and IL-23 inhibitors and highlights the scarcity of studies focusing on anogenital sites.

In addition, the use of topical corticosteroids or calcineurin inhibitors in the anogenital area may locally reduce mucosal immunity and contribute to persistent or recurrent HPV infection.

The role of biologics targeting TNF-α, IL-17, and IL-23 in the course of HPV infections therefore remains uncertain, complex, and likely dependent on immunological mechanisms that are still not fully understood. These considerations justify systematic studies to assess their specific impact on the incidence and recurrence of anogenital warts in psoriatic patients.

Finally, very limited data are available regarding risk perception of HPV infection and acceptability of HPV vaccination in this adult population receiving immunomodulatory treatments, despite the fact that prevention could be relevant.

Study Design

Type: Mixed study (retrospective + prospective) Total duration: 32 months (2025-2028) Retrospective phase: 3 months (Oct-Dec 2025) Prospective phase: 27 months (Oct/Nov 2025 - Dec 2027) Analysis phase: 5 months (Jan-May 2028)

The retrospective phase will consist of a case-control study, matching each patient who developed anogenital warts (AGW) with one or more controls receiving biologic therapy who did not develop AGW, in order to identify factors associated with their occurrence and to more precisely estimate the relative risk of AGW under biologic therapies, beyond simple case description.

Enrollment period (prospective phase): Patients will be enrolled between October and December 2025. Each patient will be followed for 24 months after enrollment, during their routine dermatology visits for psoriasis management. No additional visits will be required by the study. Relevant data will be collected during routine consultations. All data will be available prior to the start of the analysis phase.

An anonymous questionnaire on HPV vaccination acceptability will be offered during the prospective phase to all enrolled patients, regardless of vaccination status, whether or not they are receiving systemic immunomodulatory therapy (anti-TNF-α, anti-IL-17, anti-IL-23, methotrexate, cyclosporine, deucravacitinib, dimethyl fumarate). The purpose of this approach is not to promote vaccination, but to collect data on risk perception of HPV and willingness to be vaccinated, while enabling a comparative analysis between treated and untreated patients. The acceptability rate will be defined as the proportion of patients who state they would accept vaccination if it were offered.

These timelines are indicative and may be adjusted depending on the actual number of inclusions or potential delays related to ethical or logistical processes.

To ensure sufficient homogeneity in the prospective phase, both in terms of diagnosis and management, precise clinical definitions as well as a therapeutic reference document will be provided to investigators:

Anogenital wart (AGW): papillomatous lesion suggestive of HPV infection, clinically diagnosed by a dermatologist; histological confirmation may be performed in atypical or doubtful cases.

Recurrence: reappearance of lesions clinically compatible with AGW, after documented complete resolution of the initial episode.

Management of AGW will be based on French recommendations from the Haute Autorité de Santé (HAS), adapted to the Belgian therapeutic context. In particular, podophyllotoxin, recommended as first-line therapy in France, is currently unavailable in Belgium. It will therefore be replaced in the reference grid by Veregen®, which is widely used in local practice.

This adaptation is intended to guarantee a minimum level of treatment homogeneity while respecting local prescribing realities. The adapted grid will be communicated to investigators involved in the prospective phase, in order to ensure harmonization of AGW management practices during the study.

Data Collected

Common data (retrospective + prospective):

Sex, age, phototype, BMI

Type and duration of psoriasis (plaque, guttate, pustular), mode of diagnosis (clinical/histological)

Disease severity (BSA, PASI)

HPV vaccination status (vaccine, dates, and number of doses)

Current and past treatments (antipsoriatic and others, continuous or not)

Genital involvement of psoriasis: yes/no

Topical use in the genital area: molecule, duration, frequency

Comorbidities (notably HIV, diabetes, immunosuppression, chronic inflammatory diseases, etc.)

Gynecological-obstetrical status (for female patients): current pregnancy, recent pregnancy (<12 months), breastfeeding

Sexual history (relationship status, gender of sexual partners, multiple partners, unprotected intercourse, PrEP use, chemsex practices)

Addictive behaviors (smoking, drug use, alcohol)

History of STIs and anogenital warts (clinical/histological diagnosis, localization, number of lesions, dates, treatment)

History of HSIL or invasive carcinoma (cervical, anal, vulvar, vaginal, penile,

Prospective (during routine consultations):

Efficacy and adherence to antipsoriatic therapies (if patient is treated)

Occurrence/recurrence of AGW: date, localization, treatment

Occurrence/recurrence of HSIL or invasive carcinoma (cervical, anal, vulvar, vaginal, penile, or perineal)

Organization

Research nurse: administrative support

Principal investigator: recruitment, validation of inclusions, clinical supervision

Co-investigators: recruitment

Data manager: data management, anonymization, secure storage

Statistician: statistical analyses and assistance with interpretation

Statistical Analysis

Sample size calculation For the prospective phase, the power calculation was based on an expected incidence of anogenital warts (AGW) of 2% in the "topical treatments" group versus 8% in the "biologics" group (two-group design with pooled biologics; estimated distribution 50% biologics / 50% others), derived from literature data. To ensure 80% power and a two-sided alpha risk of 5%, 207 patients per group are required using either the z-test for proportions or the log-rank test (Kaplan-Meier). Allowing for a 20% loss to follow-up over 24 months, the target sample size is 498 patients in total.

For the retrospective phase, the case-control study aims to identify at least 50 cases of AGW under biologics, matched to controls at a 1:3 ratio, allowing robust multivariable analyses.

Analysis plan Analyses will be performed on an intention-to-treat basis (all enrolled patients) and per protocol (patients with at least two years of routine follow-up). Continuous variables will be described by median and interquartile range. Categorical variables will be expressed as counts and percentages.

Primary analyses

Prospective phase: Cumulative incidence of AGW will be estimated using Kaplan-Meier methods, with comparisons between treatment groups using the log-rank test. A proportional hazards Cox model will evaluate the association between treatments and risk of AGW, adjusted for the most relevant variables. The proportional hazards assumption will be checked using Schoenfeld residuals. Results will be expressed as hazard ratios with 95% confidence intervals.

Secondary analyses Predefined subgroup analyses will examine the specific effect of each therapeutic class and individual molecule.

For patients with multiple recurrences, a frailty model (a survival model designed to analyze recurrent/repeated events within individuals) will be used to account for intra-individual correlation. A sensitivity analysis excluding patients who changed treatment during follow-up will assess the robustness of the main results.

HPV vaccination acceptability will be analyzed using logistic regression, considering potential explanatory variables.

Handling of missing data Missing data will be described and their mechanism explored. If <5% of data are missing for a variable, analyses will be conducted on complete cases. For 5-20% missing data, multiple imputation using chained equations will be performed. If >20% of data are missing, the variable will be excluded from analysis.

A sensitivity analysis will compare results from complete-case and imputed datasets.

Statistical considerations To control for inflation of type I error related to multiple comparisons, the Benjamini-Hochberg procedure will be applied. The significance threshold will be set at p<0.05 after adjustment.

Analyses will be conducted using R (version 4.3 or later) or SAS (version 9.4). Results will be reported according to STROBE guidelines for observational studies, ensuring transparency and reproducibility of analyses.

Ethical Considerations

Submission to the ethics committee prior to any enrollment

Written informed consent required for the prospective phase only

GDPR compliance (anonymization, secure database, retention for 10 years)

The study does not impose any additional consultations. All data are collected exclusively during visits scheduled as part of routine clinical practice.

Appendix:

Exploratory Sub-study - Storage of Condyloma Fragments for HPV Genotyping

In certain cases, when an interventional treatment of anogenital warts (such as CO₂ laser, curettage, or other) is performed as part of routine clinical management, a small fragment may be preserved for the purpose of HPV genotyping.

These samples, collected without any additional procedure for the patient, will be stored under appropriate conditions (e.g., freezing at -80 °C or, more rarely, paraffin embedding) for possible future virological analysis in an accredited partner laboratory (likely AML Laboratory, 113 Avenue Henri Jaspar, 1160 Saint-Gilles).

The number of samples collected will depend on clinical situations encountered and technical feasibility.

This exploratory sub-study is not a primary objective of the trial but may be subject to complementary analysis if a sufficient number of samples is obtained.

This possibility has been explicitly mentioned in the patient information sheet and the informed consent form, in order to ensure transparency with participants, including in the event that no analysis is ultimately performed.

No additional costs or travel will be incurred by patients. DLQI

Perception and acceptability of HPV vaccination: specific questionnaire at baseline (M0)

Evolving gynecological-obstetrical status (for female patients): new pregnancies, current breastfeeding

Clinical examination of oral and anogenital mucosa

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Moderate to severe psoriasis (BSA > 10% or PASI > 10), prior to initiation of the current therapy at the time of inclusion
* Planned dermatological follow-up for approximately 24 months, with no additional visits required by the study
* Signed informed consent

Exclusion Criteria:

* Severe immunosuppression not related to psoriasis or its therapy (concomitant treatment with major immunosuppressants, uncontrolled HIV infection, or other conditions inducing significant immunosuppression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with moderate to severe psoriasis, not severely immunosuppressed, recruited from dermatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of anogenital warts | From enrollment until the end of the 2-year follow-up
  To evaluate the incidence of anogenital warts (AW), including both new cases and recurrences, in patients with moderate-to-severe psoriasis, by comparing major therapeutic groups: biologic therapies (anti-TNF-α, anti-IL-17, anti-IL-23, ustekinumab), other immunomodulators (methotrexate, cyclosporine, deucravacitinib, dimethyl fumarate), non-immunomodulatory systemic therapies (apremilast, acitretin), topical therapies alone (topical corticosteroids, calcineurin inhibitors, phototherapy), or no treatment.

SECONDARY OUTCOMES:
Characterization of AW cases under biologics | From enrollment until the end of the 2-year follow-up
  To identify and describe documented cases of AW in patients treated with anti-TNF-α, anti-IL-17, or anti-IL-23, analyze the circumstances of occurrence (type of biologic, time from initiation, associated factors), and assess the evolution after first appearance of AW (resolution, persistence, recurrence).
Comparison of incidence and recurrence across treatments | From enrollment until the end of the 2-year follow-up
  To compare the incidence and recurrence rates of AW across different classes or molecules of antipsoriatic treatments, including a no-treatment group, within the study cohort.
Risk factors for AW incidence and recurrence | From enrollment until the end of the 2-year follow-up
  To identify factors associated with the incidence and recurrence of AW (treatment dosage and duration, history of sexually transmitted infections, smoking, gender of sexual partners, multiple partners, unprotected sexual intercourse, and relevant comorbidities such as HIV, diabetes, or chronic inflammatory diseases).
Impact of topical genital therapies | From enrollment until the end of the 2-year follow-up
  To assess the impact of topical genital treatments (topical corticosteroids, calcineurin inhibitors), commonly used in inflammatory anogenital dermatoses, on the incidence and recurrence of AW.
HPV vaccination acceptability | At enrollment
  To evaluate the level of information and the acceptability of HPV vaccination in the entire study cohort using a structured self-administered questionnaire developed specifically for the CONDYPSO study.
  The questionnaire includes four sections (General Information, Risk Perception, Attitude Toward Vaccination, and Information Sources) composed of multiple-choice and Likert-type questions.
  Results will be analysed descriptively to assess participants' awareness, attitudes, and willingness to be vaccinated against HPV in the entire cohort, with a specific subgroup analysis among patients treated with systemic immunomodulatory therapies (anti-TNF-α, anti-IL-17, anti-IL-23, methotrexate, cyclosporine, deucravacitinib, dimethyl fumarate).
  No numerical score will be calculated; results will be presented as categorical and frequency data.
HPV genotyping in prospective cases | After completion of the 2-year follow-up of enrolled patients
  To identify the HPV genotypes involved in warts from certain patients included in the prospective phase (exploratory sub-study).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krygier, MD, Principal Investigator — CHU SAINT-PIERRE BRUXELLES
Locations (3):
- Belgium (3):
  - CHU Saint-Pierre, Brussels, Brussels Capital
  - CHU Brugmann, Brussels, Brussels Capital
  - Hôpital Erasme, Brussels, Brussels Capital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality and data protection requirements

REFERENCES:
- [Background] Karakusevic A, Foss AM. Acceptability of human papillomavirus vaccination in the United Kingdom: a systematic review of the literature on uptake of, and barriers and facilitators to HPV vaccination. Ther Adv Vaccines Immunother. 2024 Dec 25;12:25151355241308313. doi: 10.1177/25151355241308313. eCollection 2024. PMID 39737330
- [Background] Korecka K, Wisniewska-Szymanska A, Mikiel D. The impact of systemic psoriasis treatments on human papillomavirus activation and propagation. Australas J Dermatol. 2022 Aug;63(3):293-302. doi: 10.1111/ajd.13865. Epub 2022 May 4. PMID 35510323
- [Background] Burlando M, Molle MF, Cozzani E, Parodi A. Bulky Condyloma Acuminata following Ustekinumab Treatment for Plaque Psoriasis: A Case Report. Case Rep Dermatol. 2021 Apr 21;13(1):244-247. doi: 10.1159/000509178. eCollection 2021 Jan-Apr. PMID 34054460
- [Background] Avallone G, Dapavo P, Cabutti F, Preti M, Cavallo F, Roccuzzo G, Mastorino L, Rubatto M, Quaglino P, Ribero S. Regression of human papillomavirus-associated high-grade vaginal intraepithelial neoplasia after switching from ustekinumab to risankizumab in a psoriasis patient. Ital J Dermatol Venerol. 2023 Feb;158(1):61-62. doi: 10.23736/S2784-8671.22.07297-8. No abstract available. PMID 36939503
- [Background] Gosmann C, Mattarollo SR, Bridge JA, Frazer IH, Blumenthal A. IL-17 suppresses immune effector functions in human papillomavirus-associated epithelial hyperplasia. J Immunol. 2014 Sep 1;193(5):2248-57. doi: 10.4049/jimmunol.1400216. Epub 2014 Jul 25. PMID 25063870
- [Background] Walch-Ruckheim B, Stroder R, Theobald L, Pahne-Zeppenfeld J, Hegde S, Kim YJ, Bohle RM, Juhasz-Boss I, Solomayer EF, Smola S. Cervical Cancer-Instructed Stromal Fibroblasts Enhance IL23 Expression in Dendritic Cells to Support Expansion of Th17 Cells. Cancer Res. 2019 Apr 1;79(7):1573-1586. doi: 10.1158/0008-5472.CAN-18-1913. Epub 2019 Jan 29. PMID 30696656
- [Background] Sun F, Yu Z. Rapid progression of condyloma acuminatum caused by IL-17A antibody treatment: a case report. Front Med (Lausanne). 2024 May 15;11:1387620. doi: 10.3389/fmed.2024.1387620. eCollection 2024. PMID 38813385
- [Background] Kucukhemek F, Aypek Y, Ogut B, Adisen E. IL-17 Monoclonal Antibody Related HPV Exacerbation: A Case Report. Indian J Dermatol. 2024 Nov-Dec;69(6):487. doi: 10.4103/ijd.ijd_390_24. Epub 2024 Oct 29. No abstract available. PMID 39678756
- [Background] Wu DC, Salopek TG. Eruptive condyloma accuminata after initiation of infliximab treatment for folliculitis decalvans. Case Rep Dermatol Med. 2013;2013:762035. doi: 10.1155/2013/762035. Epub 2013 Dec 4. PMID 24368947
- [Background] Ferreira Torres TC, Vasconcelos Sanches M, Manuela Selores M. Development of Multiple Viral Warts in a Patient Receiving the TNF-α Inhibitor Etanercept. Psoriasis Forum. 2009;15a(2):15-6.
- [Background] Rob F, Hugo J, Salakova M, Smahelova J, Gkalpakiotis S, Bohac P, Tachezy R. Prevalence of genital and oral human papillomavirus infection among psoriasis patients on biologic therapy. Dermatol Ther. 2022 Oct;35(10):e15735. doi: 10.1111/dth.15735. Epub 2022 Aug 8. PMID 35883191
- [Background] Handisurya A, Lazar S, Papay P, Primas C, Haitel A, Horvat R, Tanew A, Vogelsang H, Kirnbauer R. Anogenital Human Papillomavirus Prevalence is Unaffected by Therapeutic Tumour Necrosis Factor-alpha Inhibition. Acta Derm Venereol. 2016 May;96(4):494-8. doi: 10.2340/00015555-2298. PMID 26581127
- [Background] Hewavisenti RV, Arena J, Ahlenstiel CL, Sasson SC. Human papillomavirus in the setting of immunodeficiency: Pathogenesis and the emergence of next-generation therapies to reduce the high associated cancer risk. Front Immunol. 2023 Mar 7;14:1112513. doi: 10.3389/fimmu.2023.1112513. eCollection 2023. PMID 36960048
- [Background] Gaffen SL, Jain R, Garg AV, Cua DJ. The IL-23-IL-17 immune axis: from mechanisms to therapeutic testing. Nat Rev Immunol. 2014 Sep;14(9):585-600. doi: 10.1038/nri3707. PMID 25145755
- [Background] Navarro-Compan V, Puig L, Vidal S, Ramirez J, Llamas-Velasco M, Fernandez-Carballido C, Almodovar R, Pinto JA, Galindez-Aguirregoikoa E, Zarco P, Joven B, Gratacos J, Juanola X, Blanco R, Arias-Santiago S, Sanz Sanz J, Queiro R, Canete JD. The paradigm of IL-23-independent production of IL-17F and IL-17A and their role in chronic inflammatory diseases. Front Immunol. 2023 Aug 4;14:1191782. doi: 10.3389/fimmu.2023.1191782. eCollection 2023. PMID 37600764
- [Background] Damiani G, Bragazzi NL, Karimkhani Aksut C, Wu D, Alicandro G, McGonagle D, Guo C, Dellavalle R, Grada A, Wong P, La Vecchia C, Tam LS, Cooper KD, Naghavi M. The Global, Regional, and National Burden of Psoriasis: Results and Insights From the Global Burden of Disease 2019 Study. Front Med (Lausanne). 2021 Dec 16;8:743180. doi: 10.3389/fmed.2021.743180. eCollection 2021. PMID 34977058
- [Background] Patel H, Wagner M, Singhal P, Kothari S. Systematic review of the incidence and prevalence of genital warts. BMC Infect Dis. 2013 Jan 25;13:39. doi: 10.1186/1471-2334-13-39. PMID 23347441
- [Background] Offidani A, Radi G, Bianchi L, Cannavo SP, Conti A, Gesuita R, Salaffi F, Talamonti M, Campanati A. Prevalence of HPV genital infection in patients with moderate-to-severe psoriasis undergoing systemic treatment with immunosuppressive agents or biologics. Eur J Dermatol. 2021 Aug 1;31(4):493-498. doi: 10.1684/ejd.2021.4121. PMID 34642139
- [Background] Al-Janabi A, Yiu ZZN. Biologics in Psoriasis: Updated Perspectives on Long-Term Safety and Risk Management. Psoriasis (Auckl). 2022 Jan 6;12:1-14. doi: 10.2147/PTT.S328575. eCollection 2022. PMID 35024352
- [Background] Ferrara F, Verduci C, Laconi E, Mangione A, Dondi C, Del Vecchio M, Carlevatti V, Zovi A, Capuozzo M, Langella R. Therapeutic Advances in Psoriasis: From Biologics to Emerging Oral Small Molecules. Antibodies (Basel). 2024 Sep 14;13(3):76. doi: 10.3390/antib13030076. PMID 39311381
- See also: HAS 2024 Guidelines on the Management of Anogenital Warts — https://www.has-sante.fr/